CLINICAL TRIAL: NCT06863519
Title: Evaluation of Endoscopic Treatment Effect and Influencing Factors in Patients With Esophageal and Gastric Varices in Cirrhosis Based on HVPG
Brief Title: Evaluation of Endoscopic Treatment Effect Based on HVPG
Status: Enrolling by invitation | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0634
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-11

CONDITIONS: Esophageal and Gastric Varices
MeSH Terms: conditions — Esophageal and Gastric Varices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic treatment — After the patient is enrolled, HVPG testing is performed, and appropriate endoscopic treatment is selected as a secondary prevention method. HVPG testing is performed again after regular endoscopic treatment.

SUMMARY:
This study aims to evaluate the endoscopic treatment effect and related influencing factors of patients with esophageal and gastric varices based on HVPG. By enrolling and collecting patients with esophageal and gastric varices at different stages of liver cirrhosis, the changes in portal pressure before and during endoscopic treatment were detected. The endoscopic treatment effect of different patients was evaluated by combining the changes in HVPG and the condition of varicose veins, the effects of different endoscopic treatment methods on HVPG were analyzed, and the correlation between HVPG changes and endoscopic efficacy was explored.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-80 years old;
2. Patients with confirmed cirrhosis through clinical, imaging or pathological evidence, with causes including viral hepatitis, alcoholic liver disease, non-alcoholic fatty liver disease, etc.;
3. Patients with esophageal and gastric varices confirmed by endoscopic examination and varicose vein bleeding in the past;
4. Endoscopic treatment (such as band ligation, sclerotherapy or colloid injection) is an appropriate secondary prevention method;

Exclusion Criteria:

* (1) Combined with hepatocellular carcinoma or other malignant tumors; (2) Autoimmune cirrhosis, schistosomal cirrhosis, hepatic venous occlusion, etc.; (3) Combined with other diseases that affect portal hypertension, such as portal vein thrombosis; (4) Recently (within 6 months) received other treatments, such as TIPS, liver transplantation, or other treatment measures that may affect the study; (5) Accompanied by severe cardiopulmonary diseases (such as severe heart failure, COPD, etc.);

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients in gastroenterology department
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
HVPG | Regular endoscopic treatment, with HVPG testing repeated approximately every 6-12 months
  After enrollment, HVPG testing was performed and appropriate endoscopic treatment was selected as a secondary prevention measure; HVPG testing was performed again approximately every 6-12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No